CLINICAL TRIAL: NCT00853606
Title: An Open-Label, Long-Term Evaluation of the Safety and Efficacy of Avanafil in Men With Erectile Dysfunction
Brief Title: Long-Term Safety and Efficacy Study of Avanafil in Men With Erectile Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TA-314
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Results first posted 2012-06-28 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Erectile Dysfunction
Keywords: ED; Erectile Dysfunction; Dysfunction; Erectile
MeSH Terms: conditions — Erectile Dysfunction | interventions — avanafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- avanafil (Experimental)
  Interventions: Drug: avanafil

INTERVENTIONS:
Drug: avanafil — All subjects will initially be assigned to treatment with avanafil 100 mg. Subjects who are unable to tolerate treatment with 100 mg may undergo dose reduction to 50 mg. Subjects who tolerate avanafil 100 mg but who desire increased efficacy may request a dose increase to 200 mg.
  Other Names: TA-1790; Stendra

SUMMARY:
This open-label study is being conducted to evaluate the long-term safety, tolerability, and efficacy of avanafil in men with mild to severe erectile dysfunction. Approximately 400 subjects will be enrolled and treated with avanafil for up to 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Successfully completed the entire treatment period in a qualifying study (TA-301 [NCT00790751] or TA-302 [NCT00809471]);
* Demonstrated compliance with the study protocol, including drug administration, diary completion, and scheduled study visits, during the qualifying trial;
* Made at least 4 attempts at intercourse during the last treatment period of the qualifying trial;
* Agree to make at least 4 attempts at intercourse each month through the course of this study;
* Agree not to use any other treatments for erectile dysfunction during participation in this study.
* Provide written informed consent;
* Willing and able to comply with scheduled study visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Subjects who, in the opinion of the investigator, have developed one or more comorbidities during the qualifying study that would pose a safety concern to their continuation on treatment in study TA-314;
* Subjects requiring treatment with an excluded medication.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 712 (Actual)
Dates: Start 2009-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McCullough, MD, Principal Investigator — NYU Urology Associates
Locations (37):
- United States (37):
  - Research Site, Birmingham, Alabama
  - Research Site, Homewood, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Waterbury, Connecticut
  - Research Site, Clearwater, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jupiter, Florida
  - Research Site, Ocala, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Ponte Vedra, Florida
  - Research Site, Tampa, Florida
  - Research Site, Sandy Springs, Georgia
  - Research Site, Wichita, Kansas
  - Research Site, Madisonville, Kentucky
  - Research Site, Shreveport, Louisiana
  - Research Site, Kansas City, Missouri
  - Research Site, Lawrenceville, New Jersey
  - Research Site, Albany, New York
  - Research Site, New York, New York
  - Research Site, Cary, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Harrisburg, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Bala-Cynwyd, Pennsylvania
  - Research Site, Lancaster, Pennsylvania
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, Spring, Texas

REFERENCES:
- [Derived] Belkoff LH, McCullough A, Goldstein I, Jones L, Bowden CH, DiDonato K, Trask B, Day WW. An open-label, long-term evaluation of the safety, efficacy and tolerability of avanafil in male patients with mild to severe erectile dysfunction. Int J Clin Pract. 2013 Apr;67(4):333-41. doi: 10.1111/ijcp.12065. PMID 23521325

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment occurred at US investigative sites between March 2009 and April 2010.
Groups:
- Avanafil: All subjects will initially be assigned to treatment with avanafil 100 mg. Subjects who are unable to tolerate treatment with the 100 mg dose may request a dose reduction to 50 mg. Study medication should be taken orally with water 30 minutes prior to the initiation of sexual activity.
Period: Overall Study
Arm/Group | Avanafil
Started | 712
Completed | 492
Not Completed | 220

BASELINE CHARACTERISTICS:
Arm/Group | Avanafil
Number analyzed (Participants) | 712
Age Continuous [Mean (Standard Deviation); unit: years] | 56.4 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 712
Region of Enrollment [Number; unit: participants]
  United States | 712

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage of Sexual Attempts in Which Subjects Were Able to Maintain an Erection of Sufficient Duration to Have Successful Intercourse.
Description: Data presented as mean change from baseline and the treatment period in the percentage of Yes responses to Sexual Encounter Profile (SEP) diary question 3 "Did your erection last long enough for you to have successful intercourse?" Baseline is the run-in period from the qualifying study (TA-301/TA-302) consisting of all data reported during the non-treatment interval from Visit 1 to Visit 2. The treatment period is the on-treatment interval beginning with the first dose of study drug and ending on the last study visit.
Time Frame: Baseline, 52 weeks
Population: Number of participants analyzed represents the Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: percentage of sexual attempts
Arm/Group | Avanafil
Number analyzed (Participants) | 686
percentage of sexual attempts | 54.75 (35.915)

2. Primary Outcome: Change in Percentage of Sexual Attempts in Which Subjects Were Able to Insert the Penis Into the Partner's Vagina
Description: Data presented as mean change from baseline and the treatment period in the percentage of Yes responses to Sexual Encounter Profile (SEP) diary question 2 "Were you able to insert your penis into your partner's vagina?" Baseline is the run-in period from the qualifying study (TA-301/TA-302) consisting of all data reported during the non-treatment interval from Visit 1 to Visit 2. The treatment period is the on-treatment interval beginning with the first dose of study drug and ending on the last study visit.
Time Frame: Baseline, 52 weeks
Population: Number of participants analyzed represents to Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: percentage of sexual attempts
Arm/Group | Avanafil
Number analyzed (Participants) | 686
percentage of sexual attempts | 36.91 (36.142)

3. Primary Outcome: Change in International Index of Erectile Function - Erectile Function Domain (IIEF-EF) Score
Description: Questionnaire assesses subject's evaluation of erectile function over the previous 4-week period. Total score from questions 1-5 & 15 ranges from 1 to 30. A higher score indicates better erectile function. Baseline is the observation at Visit 2 of the qualifying study (TA-301/TA-302). End of treatment is the observation at Visit 8 of the last observation carried forward.
Time Frame: Baseline, End of Treatment
Population: Number of participants analyzed represents the Intent-to-Treat population. For dropouts of missing data, the last observation carried forward convention was used.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Avanafil
Number analyzed (Participants) | 686
scores on a scale | 10.3 (7.88)

ADVERSE EVENTS:
Time Frame: AE reporting began when the subject provided written informed consent and extended until 28 calendar days after the last dose of the investigational product was administered, or until the subject was discontinued from the study, whichever was later.
Description: # participants at risk is presented for the safety population. The Safety Population was defined as all subjects who received at least one dose of avanafil during TA-314 and who have any safety data.
Arm/Group | Avanafil
Serious Adverse Events (participants affected / at risk) | 11/712
Other Adverse Events (participants affected / at risk) | 87/712
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avanafil (N=712)
Acute physchosis (Psychiatric disorders) | 1
pancreatitis acute (Gastrointestinal disorders) | 1
femoral artery occlusion (Vascular disorders) | 1
inguinal hernia (Gastrointestinal disorders) | 1
syncope vasovagal (Nervous system disorders) | 1
coronary artery disease (Cardiac disorders) | 1
cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
subdural hematoma (Injury, poisoning and procedural complications) | 1
atrial fibrillation (Cardiac disorders) | 1
aortic valve stenosis (Cardiac disorders) | 1
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
small intestinal obstruction (Gastrointestinal disorders) | 1
cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
cardiac failure congestive (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avanafil (N=712)
nasopharyngitis (Infections and infestations) | 24
headache (Nervous system disorders) | 40
flushing (Vascular disorders) | 25
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After Sponsor's written notification that publication of results is no longer planned or 12 months after termination of the study at all sites, Institution & PI may publish, upon written approval from Sponsor, results of the Study. Sponsor will be given the opportunity to review any proposed publication at least 60 days prior to submission for publication or disclosure. Upon Sponsor's written request, Institution and PI shall not publish or disclose information related to the Study.